CLINICAL TRIAL: NCT06386211
Title: Open-label, Randomized, 2-treatment, 2-sequence, 2-period, Crossover Relative Bioavailability Study of Magne-B6 New Formulation Versus Magne-B6 Solution in Healthy Male and Female Subjects in Fasting Conditions.
Brief Title: Bioavailability Study of Magne-B6 New Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opella Healthcare Group SAS, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDR17228; BDR17228 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence Group 1 (Experimental)
  Interventions: Drug: MAGNE-B6 Oral Solution; Drug: MAGNE-B6 New Formulation Tablet
- Treatment Sequence Group 2 (Experimental)
  Interventions: Drug: MAGNE-B6 Oral Solution; Drug: MAGNE-B6 New Formulation Tablet

INTERVENTIONS:
Drug: MAGNE-B6 Oral Solution — Oral solution.
Drug: MAGNE-B6 New Formulation Tablet — New formulation tablet.

SUMMARY:
The purpose of the study is to assess the relative bioavailability of two Magne-B6 preparations, in fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, between 18 and 45 years of age, inclusive.
2. Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive.
3. Females of childbearing potential (pre-menopausal female biologically capable of becoming pregnant) or not documented post-menopausal (menopause is defined as being amenorrheic for at least 1 year with plasma follicle stimulating hormone [FSH] level >30 International units per liter [UI/L]) who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last IMP administration:

   * Intra-uterine contraceptive device placed at least 4 weeks prior to IMP administration.
   * Male condom with intravaginally applied spermicide starting at least 21 days prior to investigational medicinal product (IMP) administration.
   * Hormonal contraceptives starting at least 4 weeks prior to IMP administration and must agree to use the same hormonal contraceptive throughout the study.
   * Sterile male partner (vasectomized since at least 6 months).
   * Abstaining from sexual intercourse.
4. Male participant, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, an adequate contraception for study period duration or abstaining from sexual intercourse.
5. Presenting normal magnesemia (0.65-1.05 millimolar [mM]).
6. Presenting normal plasma level of vitamin B6 (20-50 nanomolar [nM]).
7. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
8. Vital signs after 10 minutes resting in supine position within the following range:

   * Systolic blood pressure (SBP): 100 - 130 millimeters of mercury (mmHg)
   * Diastolic blood pressure (DBP): 60 - 90 mmHg
   * Heart rate (HR): 60 -90 beats per minute (bpm).
9. Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges: 120 milliseconds (ms)<PQ<200 ms, 60 ms <QRS<100 ms, QTcF from 340 ms to 450 ms inclusive and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
10. Laboratory parameters within the normal range.
11. Having given written informed consent prior to undertaking any study-related procedure.
12. Not under any administrative or legal supervision

Exclusion Criteria:

1. Lactase deficiency, lactose intolerance; glucose-galactose malabsorption; acute infectious diseases or allergic reaction requiring treatment (including drug allergies) within 4 weeks prior to the screening; a history of gastrointestinal tract surgery (except appendectomy).
2. Depot injections, installation of intrauterine hormonal therapeutic systems or implants of any drugs 6 months before the first day of screening.
3. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
4. Participants experiencing stress, especially severe stress, anxiety, post-trauma or social anxiety disorder, or depression would be excluded.
5. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
6. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
7. Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
8. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
9. For women: using hormonal contraceptives less than 2 months before the first day of screening.
10. Participants receiving hormonal replacement therapy (incl. surgical menopause).
11. Any medication, vitamin, biologically active additives, herbal preparations (including St John's Wort, angelica, evening primrose, feverfew, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng, etc.) within 30 days before inclusion any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before screening.
12. Any intake of aluminum-and-magnesium-containing antacids within 14 days before Period I.
13. Any drug containing Magnesium or B6 vitamin within 14 days before Period I.
14. Any tricyclic antidepressants within 14 days before Period I.
15. Deviations of laboratory test results from reference intervals standard laboratory and instrumental examination methods.
16. Any diet, such as vegetarian, within 2 weeks of the first day of screening.
17. Not being able to go without food for at least 12 hours and not being able to take the drug on an empty stomach.
18. Volunteers expected to have problems with venous catheterization or venipuncture.
19. Volunteers unwilling or unable to give up alcohol and excessive exercise from the first day of screening to the follow-up visit.
20. Volunteers with lifestyles (including night work and extreme physical activity such as sports or weightlifting) that can make it difficult to interpret laboratory findings from the study.
21. Volunteers who are unwilling to observe the requirements of the study and / or unreliable, volunteers who, in the Investigator's opinion, are apparently or probably unable to understand and assess information concerning this study before the signing of the Informed Consent Form, in particular in relation to anticipated risks and potential discomforts.
22. Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
23. Participation in any other clinical trial or study drug intake less than 3 months before the first day of screening.
24. Any participant who cannot be contacted in case of emergency.
25. Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
26. Any consumption of citrus fruits (grapefruit, orange, etc.) or their juices, as well as all fruit juices, within 5 days before Period I.
27. Alcohol consumption more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse.
28. Smoking regularly more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
29. Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
30. If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-HCG] blood test), or breast-feeding.
31. Premenstrual syndrome
32. Climacteric syndrome (incl. surgical menopause) not receiving hormonal replacement therapy.
33. Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus antibodies (anti-HIV Ab).
34. Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
35. Positive alcohol breath test.
36. Presence or history of hypersensitivity to any presentation of Magne-B6 or to any of the excipients.
37. Participants presenting one or several symptoms of magnesium deficiencies as listed in the Magne-B6 summary of product characteristic (SmPC).
38. Any contraindications to Magne-B6, according to the applicable labeling.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Maximal Observed Concentration (Cmax) of Magnesium in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Area Under the Concentration-time Curve from Time Zero Until time 12 hour (h) (AUC0-12) of Magnesium in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Area Under the Concentration-time Curve from Time Zero Until time 24 h (AUC0-24) of Magnesium in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Maximal Observed Concentration (Cmax) of Pyridoxine in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Area Under the Concentration-time Curve from Time Zero Until the Last Observed Concentration (AUClast) of Pyridoxine in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Area Under the Concentration-time Curve from Time Zero to Infinity (extrapolated) (AUC0-infinity) of Pyridoxine in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Time When the Maximal Concentration is Observed (Tmax) of Magnesium in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Time When the Maximal Concentration is Observed (Tmax) of Pyridoxine in Plasma | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2
Cumulative Amount of Unchanged Drug Excreted into the Urine From Time Zero to the Time Point 24 hours (Ae0-24) of Magnesium in Urine | Pre-dose and Days 1 and 2 after the treatment administration in Period 1 and 2

SECONDARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | From screening up to 3 days after last administration (approximately 7 weeks)
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical trial participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment.
  A TEAE is defined as an AE that occurred or worsened at any time during the on-treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: CHC Clinical studies, Study Director — Opella Healthcare Group SAS, a Sanofi Company
Locations (1):
- Erciyes Universitesi Hakan Cetinsaya Iyi Klinik Uygulama ve Araştırma Merkezi Erciyes Universitesi Kampusu, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BDR17228 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26031&tenant=MT_SNY_9011